CLINICAL TRIAL: NCT00503594
Title: Multicenter Randomized Phase II Study of Methotrexate (MTX) and Temozolomide Versus MTX, Procarbazine, Vincristine and Cytarabine for Primary CNS Lymphoma (PCNSL) in the Elderly
Brief Title: Methotrexate and Temozolomide Versus Methotrexate, Procarbazine, Vincristine and Cytarabine
Acronym: CNSLymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060239
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Lymphoma
Keywords: Primary central nervous system lymphoma; Brain lymphoma; Elderly; Chemotherapy; Methotrexate; Temozolomide; Procarbazine; Vincristine; Cytarabine
MeSH Terms: conditions — Lymphoma | interventions — Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Comparative evaluation of the efficiency of a new protocol of the primitive LYMPHOME of the central nervous system ( LPSNC) to the old subject, associating Methotrexate and Temozolomide with regard to a standard protocol associating Methotrexate, Procarbazine, Vincristine and Cytarabine.
  Interventions: Drug: Methotrexate and temozolomide
- bras conventional (Active Comparator): bras conventional
  Interventions: Drug: Methotrexate , procarbazine ,vincristine ,cytarabine

INTERVENTIONS:
Drug: Methotrexate and temozolomide — Methotrexate and temozolomide
  Arms: 1
Drug: Methotrexate , procarbazine ,vincristine ,cytarabine — Methotrexate , procarbazine ,vincristine ,cytarabine
  Arms: bras conventional

SUMMARY:
The purpose of this study is to evaluate two types of chemotherapy for primary central nervous system lymphoma in the elderly (age older than 60) :

* Methotrexate, procarbazine, vincristine and cytarabine
* Methotrexate and temozolomide

DETAILED DESCRIPTION:
The aim of the study is to evaluate efficacy and toxicity associated with both protocols in this population, without radiotherapy.

Patients will be randomized to receive one of the two regimens in one of the participating centers. Neuropsychological evaluation will be performed in all patients. Patients will be followed with serial MRIs.

ELIGIBILITY:
Inclusion Criteria:

* primary central nervous system lymphoma histologically confirmed by brain biopsy, CSF cytology or vitrectomy
* KPS 40 or higher
* Absence of systemic disease as evaluated by chest-abdomen-pelvis CT scan
* Leucocytes>3.500/mm3, platelets>130.000/mm3, Bilirubin < 2 mg, transaminases < 2.5 N), creatinine < 150 μM/l, creatinine clearance > 40 ml/min
* Age ≥ 60 years
* Negative HIV test
* Signature of informed consent

Exclusion Criteria:

* previous cranial radiotherapy
* prior chemotherapy for primary central nervous system lymphoma
* presence of another cancer (excepting basal cell carcinoma of the skin and cervical carcinoma in situ )
* systemic lymphoma (outside the CNS)
* Isolated ocular lymphoma
* Immunosuppressed patients (HIV , use of immunosuppressors)
* Other uncontrolled or progressive disease compromising shot-term survival
* Severe renal or hepatic disease
* Patients not legally covered by the French Social Security
* Inability to swallow the medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | at one year

SECONDARY OUTCOMES:
Overall survival:median and overall survival | at one and two years
Response rates | at end of treatment
Toxicity | during treatment
Late toxicity | 2 to 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio OMURO, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe hospitalier la Pitié Salpétrière, Paris, France

REFERENCES:
- [Result] Omuro AM, Abrey LE. Chemotherapy for primary central nervous system lymphoma. Neurosurg Focus. 2006 Nov 15;21(5):E12. doi: 10.3171/foc.2006.21.5.13. PMID 17134114
- [Derived] Omuro A, Chinot O, Taillandier L, Ghesquieres H, Soussain C, Delwail V, Lamy T, Gressin R, Choquet S, Soubeyran P, Huchet A, Benouaich-Amiel A, Lebouvier-Sadot S, Gyan E, Touitou V, Barrie M, del Rio MS, Gonzalez-Aguilar A, Houillier C, Delgadillo D, Lacomblez L, Tanguy ML, Hoang-Xuan K. Methotrexate and temozolomide versus methotrexate, procarbazine, vincristine, and cytarabine for primary CNS lymphoma in an elderly population: an intergroup ANOCEF-GOELAMS randomised phase 2 trial. Lancet Haematol. 2015 Jun;2(6):e251-9. doi: 10.1016/S2352-3026(15)00074-5. Epub 2015 Jun 3. PMID 26688235
- See also: A review on chemotherapy options for primary central nervous system lymphoma — http://www.ncbi.nlm.nih.gov